CLINICAL TRIAL: NCT06639997
Title: A Phase I Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AZD5148 in Healthy Japanese Adults
Brief Title: Safety and Tolerability of AZD5148 in Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D8820C00005
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Clostridioides Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 - AZD5148 IM (Experimental): Biological: AZD5148 (Cohort 1)
  ・Single dose of AZD5148 IM
  Interventions: Drug: AZD5148
- Cohort 1 - Placebo IM (Placebo Comparator): Biological: Placebo (Cohort 1) Single dose of Placebo IM
  Interventions: Drug: Placebo
- Cohort 2 - AZD5148 IV (Experimental): Biological: AZD5148 (Cohort 2)
  ・Single dose of AZD5148 IV
  Interventions: Drug: AZD5148
- Cohort 2 - Placebo IV (Placebo Comparator): Biological: Placebo (Cohort 2) Single dose of Placebo IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD5148 — Participants will receive AZD5148 as IM injection or IV bolus
  Arms: Cohort 1 - AZD5148 IM; Cohort 2 - AZD5148 IV
Drug: Placebo — Participants will receive matching doses of placebo as an IM injection or IV bolus
  Arms: Cohort 1 - Placebo IM; Cohort 2 - Placebo IV

SUMMARY:
The purpose of this study is to measure safety, tolerability and PK of a single dose of AZD5148 administered via IV bolus or IM injection in healthy Japanese participants.

DETAILED DESCRIPTION:
The purpose of this study is to measure safety, tolerability and PK of a single dose of AZD5148 administered via IV bolus or IM injection in healthy Japanese participants.

Study details include:

• There will be 12 planned visits (including screening visit) over a period of up to 56 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be Japanese male or female and aged 18-65 years inclusive at the time of signing the informed consent.
* Participants who are overtly healthy, as determined by medical evaluation, including medical history, physical examination and baseline safety laboratory studies, according to the judgement of the investigator.
* Electrocardiograms without clinically significant abnormalities at screening.
* Able to complete the Follow-up Period through Day 361 as required by the protocol.
* No medical history of symptomatic C. difficile infection within the prior 2 years.
* Participants must be medically stable, defined as disease not requiring significant change in therapy or hospitalisation or worsening disease during the 1 month prior to enrolment, with no acute change in condition at the time of study enrolment as judged by the Investigator.
* Able to understand and comply with study requirements/procedures based on the assessment of the Investigator.
* Body weight within the range of 45 to 110 kg and body mass index (BMI) within the range of 18.0 to 32.0 kg/m2 (inclusive) at screening.
* Contraceptive use by women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Women of no childbearing potential are defined as women who are either permanently sterilised or postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to the planned date of randomisation without an alternative medical cause. The following age-specific requirements apply:

     * Women < 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following the cessation of exogenous hormonal treatment and follicle-stimulating hormone levels in the postmenopausal range.
     * Women ≥ 50 years old would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following the cessation of all exogenous hormonal treatment.
  2. Female participants of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. Women of childbearing potential who are sexually active with a non-sterilised male partner must agree to use one highly effective method of birth control from 3 months prior to IMP administration and agree to continue through 360 days following IMP administration. Cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, withdrawal, spermicides only and lactational amenorrhoea method are not acceptable methods of contraception. Female condom and male condom should not be used together. All women of childbearing potential must have negative results of pregnancy tests prior to dosing.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Previous hypersensitivity, infusion-related reaction or severe adverse reaction following mAb administration.
* Abnormal vital signs after 5 minutes of supine rest, at Screening and/or admission to the study site.
* Any clinically important abnormalities in laboratory values at the Screening Visit.
* Clinically significant bleeding disorder or prior history of significant bleeding or bruising following IM injections or venipuncture
* Primary or acquired immunodeficiency, including HIV infection, or due to drugs, including any course of glucocorticoid therapy exceeding 2 weeks of prednisone or equivalent at a dose of 20 mg daily or every other day within 6 months prior to screening. Any known HIV infection at screening
* Any known hepatitis B or C virus infection at screening
* History of malignancy other than treated non-melanoma skin cancers or locally treated cervical cancer in the previous 5 years
* Any laboratory value in the screening panel that, in the opinion of the investigator, is clinically significant or might confound analysis of study results
* Absence of suitable veins for blood sampling and IMP administration
* Receipt of immunoglobulin or blood products, or expected receipt, within 6 months prior to screening or expected to receive during the study
* Previous receipt of an mAb within 6 months or five antibody half-lives (whichever is longer), prior to informed consent date
* Receipt of any investigational products in the preceding 90 days or expected receipt of investigational product during the period of study follow-up or concurrent participation in another interventional study
* Participants with a known hypersensitivity to any component of the IMP
* History of allergic disease or reactions likely to be exacerbated by any component of the IMP
* Blood drawn in excess of a total of 400 mL (1 unit) for any reason within 3 months prior to screening or plan to donate blood until the end of follow-up period
* History of alcohol or drug abuse within the past 2 years that, according to the investigator, might affect the assessments of safety or ability the of participant to comply with all study requirements
* Deprived of freedom by an administrative or court order, in an emergency setting or hospitalised involuntarily
* Any condition that, in the opinion of the investigator, might compromise participant safety or interfere with the evaluation of the IMP or interpretation of participant safety or study results. The investigator should follow the standard vital sign ranges
* Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restriction sand requirements.
* Previous randomisation in the present study.
* For females only - currently pregnant or breast-feeding.
* Employees of the sponsor, study site or any other individuals involved with the conduct of the study or immediate family members of such individuals.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Number of Japanese participants with adverse events (AEs). | From Randomization (Day -1 or Day 1) to Day 91
  To evaluate the safety and tolerability of AZD5148 administered as a single IV or IM dose to healthy Japanese adult participants.
Number of participants with serious adverse events (SAEs) | From Screening (Day -28 to Day -2) to final Follow-up Visit (Day 361)
  To evaluate the safety and tolerability of AZD5148 administered as a single IV or IM dose to healthy Japanese adult participants.
Number of participants with adverse events of special interest (AESIs) | From Randomization (Day -1 or Day 1) to final Follow-up Visit (Day 361)
  To evaluate the safety and tolerability of AZD5148 administered as a single IV or IM dose to healthy Japanese adult participants.

SECONDARY OUTCOMES:
Maximum observed drug concentration (Cmax) | From Day 1 until last Follow up visit (Day 361)
  To evaluate the single dose PK of AZD5148.
Time to reach maximum observed concentration (tmax) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Time of last quantifiable concentration (tlast) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Terminal elimination half-life, estimated as (ln2)/λz (t1/2λz) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Area under concentration-curve from time 0 to the time of last quantifiable concentration (AUClast) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Area under concentration-time curve from time 0 extrapolated to infinity (AUCinf) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Volume of distribution at steady state (IV administration only) (Vss) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Volume of distribution at terminal phase (IV administration only) (Vz) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Systematic clearance (IV administration only) (CL) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Apparent total body clearance (IM administration only) (CL/F) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Apparent volume of distribution based on the terminal phase (IM administration only) (Vz/F) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Bioavailability for extravascular administration (IM administration only) (F) | From Day 1 until last Follow up visit (Day 361 days)
  To evaluate the single dose PK of AZD5148.
Incidence of positive ADAs against AZD5148 in serum | Day 1 (pre-dose), Day 29, Day 91, Day 181 and Day 361
  To evaluate the ADA responses to a single IV or IM dose of AZD5148.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/